CLINICAL TRIAL: NCT02983734
Title: D-cycloserine: A Novel Treatment for Gulf War Illness
Brief Title: D-cycloserine: A Novel Treatment for Gulf War Illness (GWDCS)
Acronym: GWDCS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, RosemaryToomey, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-15-1-0588
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Gulf War Illness
Keywords: Gulf War; D-cycloserine; Neuroinflammation; Cognition; Memory
MeSH Terms: conditions — Neuroinflammatory Diseases | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Active Comparator): To compare efficacy of the novel therapeutic approach of DCS in improving cognitive functioning in GW veterans with GWI.
  DCS = d-cycloserine
  Dosage: 100mg
  Dosage form: Pill, administered orally
  Frequency: Daily for four weeks
  Interventions: Drug: D-cycloserine
- Placebos (Placebo Comparator): To provide a control group to compare efficacy of the novel therapeutic approach of DCS in improving cognitive functioning in GW veterans with GWI.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: D-cycloserine — Partial agonist of N-methyl-D-aspartate (NMDA) receptor
  Other Names: DCS
  Arms: D-cycloserine
Drug: Placebos — Sugar pill
  Other Names: Placebo control
  Arms: Placebos

SUMMARY:
The purpose of this study is to investigate the efficacy of d-cycloserine (DCS) treatment for Gulf War Illness (GWI). Gulf War veterans with Gulf War Illness experience numerous chronic health symptoms, including cognition and fatigue, which reduces their quality of life. Gulf War veterans are in urgent need of novel treatment plans to tackle elusive symptomatology of Gulf War Illness. By using the literature of previous studies, the investigators have chosen to investigate d-cycloserine as a possible candidate for treating GWI, specifically cognitive symptoms. DCS has been shown to reduce neuroinflammation, regulate glutamate levels, and improve synaptic functioning in key areas of the brain.

DETAILED DESCRIPTION:
Our study is a pilot study for the novel treatment of d-cycloserine to treat GWI. Our study will consist of two experimental groups of equal size (n=28): DCS treatment group and a placebo group. Participants will be randomized into either group; with a double blind study design. Participants will be instructed to self-administer their treatment pills once per day for 28 days. There will be a total of 6 study visits that will include medical and neuropsychological assessment. The first visit will be for establishing eligibility and baseline functioning. Three visits (visits 2-4) will occur during the medication trial (day 1, day 2 and two weeks into medication/placebo). Visit 5 will occur around the time medication/placebo is finished. Visit 6 (follow up) will occur one month after medication/placebo is complete.

ELIGIBILITY:
Inclusion Criteria:

* Veterans of the 1991 Gulf War, male or female
* Physical examination and laboratory findings within normal limits
* Willingness and ability to participate in the informed consent process and comply with study protocols
* Symptom criteria: Meets Gulf War Illness criteria with the cognitive symptom domain being present. Veteran does not have medical exclusions for Gulf War Illness

Exclusion Criteria:

* Veteran lacks the capacity to provide consent during the informed consent process
* Veteran has the one of the following medical exclusion conditions and/or has been active or received treatment within the past 5 years: Cancer (except nonmelanoma skin cancer), diabetes (not well managed), seizure disorder, heart disease (except hypertension), liver disease, kidney disease, Lupus, multiple sclerosis, stroke, chronic infectious disease, immune disorder/immunosuppression
* Veteran has a history of a major psychiatric or central nervous system disorder that can affect cognitive function (ie. epilepsy, brain tumor, Parkinson's Disease)
* Veteran has been hospitalized in the past 5 years for depression, PTSD, alcohol or drug dependence
* Veteran has current suicidal ideation or current alcohol or drug dependence
* Pregnant women, lactating women, women who are breastfeeding, or women of childbearing potential who are not using medically accepted forms of contraception
* Veteran is active duty personnel

Ages: 43 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Test Battery | 8 weeks per subject

SECONDARY OUTCOMES:
Symptom Questionnaires | 8 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Toomey, Ph.D., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No